CLINICAL TRIAL: NCT05449743
Title: Evaluation of the Effectiveness of a Phlebology-oriented Spa Treatment on the Quality of Life of Patients Suffering from Chronic Venous Insufficiency of the Lower Limbs, 6-month After the Spa Treatment
Brief Title: Assessment of the Effect of Spa Therapy on the Quality of Life of Patients with Chronic Venous Insufficiency (NEYRAC)
Acronym: NEYRAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Le Syndicat Intercommunal pour le Thermalisme et l'Environnement (Other)
Collaborators: Floralis (Industry); University Grenoble Alps (Other); thermes de NEYRAC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-A00545-36
Record Dates: First submitted 2022-06-23; First posted 2022-07-08 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Chronic Venous Insufficiency
Keywords: spa therapy; phlebology; chronic venous insufficiency

STUDY DESIGN:
Intervention Model Description: before / after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patient treated with a phlebology-oriented spa therapy (Experimental): Thermal treatments among the following: pool, Kneipp pool, high pressure shower under immersion in a swimming pool, general jet shower, cataplasm in multiple local application, compress, massage under water or with thermal derivatives, walking corridor
  Interventions: Other: Spa therapy

INTERVENTIONS:
Other: Spa therapy — Thermal treatments among the following: pool, Kneipp pool, high pressure shower under immersion in a swimming pool, general jet shower, cataplasm in multiple local application, compress, massage under water or with thermal derivatives, walking corridor
  Other Names: spa treatment; spa care

SUMMARY:
Evaluation of the effectiveness of a phlebology-oriented spa therapy at 6 months on the quality of life of patients suffering from chronic venous insufficiency of the lower limbs

DETAILED DESCRIPTION:
NEYRAC is a:

* prospective, before/after, cohort follow-up study with repeated measurements
* monocentric study with the dispensation of a 3-week phlebology-oriented spa therapy in Neyrac-les-Bains

ELIGIBILITY:
Inclusion criteria:

* Age greater than 18 years
* Patient with chronic venous insufficiency of the lower limbs (CEAP category C4a, C4b and C4c)
* Patient presenting an indication for a phlebology-oriented spa treatment as the primary orientation. Patients with a dermatological or rheumatological pathology can benefit from a dual orientation spa treatment with a main phlebology orientation
* Patient affiliated to the social security system or such a system
* Available for an 18-day spa treatment and a 6-month follow-up
* For women of childbearing age: effective contraception
* Patient close to a study investigator (excluding teleconsultation) If not patient with access to the necessary equipment to perform a teleconsultation (smartphone, tablet or computer with an internet connection + taking and sending photos of the lower limbs)

Non inclusion criteria:

* Venous surgery or venous interventional therapy within 3 months prior to inclusion or scheduled within the next 3 months
* History of venous ulcer
* Contraindication to spa therapy (immune deficiency, evolving cardiopathy neoplasia, infection, pulmonary tuberculosis, severe renal insufficiency, alcoholic cirrhosis, advanced senility and severe mental disorders)
* Predictable intolerance to thermal treatments (intolerance to heat, baths, etc.)
* Persons suffering from venous insufficiency of the varicose vein type (category CEAP C2) or edema alone (category CEAP C3) or open or healed ulcers (CEAP category C5 and C6)
* Patient who has already undergone a phlebology-oriented spa treatment within the current thermal season
* Subject already included in an interventional clinical research protocol
* Persons referred to in articles L1121-5 to L1121-8 of the "Code de la Santé Publique" (pregnant women, women in labour and parturient and nursing mothers, persons deprived of liberty by judicial or administrative decision, persons subject to a legal protection measure or not being able to verbally communicate their agreement, minor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of a complete phlebology-oriented spa therapy on the quality of life of patients suffering from chronic venous insufficiency of the lower limbs | 6 months
  Comparison of the mean scores of the Chronic Venous Insufficiency specific Quality of life questionnaire (CIVIQ20) at baseline and at 6 months.
  The 20-item questionnaire, which provides a global index and an outline of 4 quality-of-life dimensions-"pain" (4 items), "physical" (4 items), "psychological" (9 items), and "social" (3 items).
  Items on the CIVIQ-20 scale were scored from 1 to 5 which means a total score from 20 to 100.
  A higher score means a worse outcome.

SECONDARY OUTCOMES:
Comparison of Visual Analog Scales (VAS) for pain at enrolment and 1.5, 3, 4.5 and 6 months after enrolment (post-cure) to quantitatively assess the improvement of patients' pain before/after treatment | 1.5, 3, 4.5 and 6 months
  Comparison of the means of Visual Analog Scales (VAS) at enrolment an 1.5, 3, 4.5 and 6 months after enrolment.
  Score from 0 to 100. A higher score means a worse outcome.
Assessment of the global quality of life by the EuroQol 5 Dimensions 5 Levels questionnaire (EQ5D-5L). | 3 and 6 months
  Improvement in global quality of life (EQ5D-5L questionnaire) between enrolment and at 3 and 6 months after enrolment
  The EQ5D-5L essentially consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  There are five dimensions assessed in the descriptive system: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  Score from -0.53 to 1. A higher score means better outcome.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
  Score from 0 to 100. A higher score means better outcome.
Physician/Patient perception | 3 and 6 months
  The perception of the physician and the patient will be asked to evaluate the benefit of the spa therapy, 3 and 6 months after enrolment using a 5-point Likert scale.
  There are no numerical scores, only results in % of patients improved or worsened.
Medication consumption | 6 months
  Collection of medication consumption to evaluate the benefit of the spa therapy (comparison of consumption before and after treatment)
  To avoid any risk of confusion, medication consumption will be set to the daily consumption. Medication use for 72 hours (D-2, D-1, D0)
  Medication consumption day before yesterday/yesterday/today:
  * Anticoagulant
  * Veinotonic
  In the 3 months prior to the visit:
  Medication use will be assessed by the investigating physician who will have to specify if this one is consumed because of the venous insufficiency or of another pathology
Assessment of compression compliance | 3 and 6 months
  Comparison of the self-reported compression compliance (percentage of wearing time in the last week), between baseline and 3 and 6 months after enrolment
Evolution of the CEAP (Clinical Etiology Anatomical distribution Pathophysiology) category | 3 and 6 months
  Comparison of CEAP category assessed by the investigating physician between enrolment and 3 and 6 months after enrolment
  The basic principles of the CEAP classification include a description of the clinical class (C) based on objective signs, the etiology (E), the anatomical distribution (A) of reflux and obstructions in superficial, deep and perforating veins and the underlying pathophysiology (P), whether related to reflux or obstructions.
  Only the clinical class (C) and the etiology (E) will be assessed.
Evolution of the general clinical criteria : Body Mass Index (BMI) | 3 and 6 months
  Comparison of the Body Mass Index between enrolment, and 3 months and 6 months after enrolment
Evolution of the general clinical criteria : systolic blood pressure | 3 and 6 months
  Comparison of the systolic blood pressure between enrolment, and 3 months and 6 months after enrolment
Evolution of the general clinical criteria : diastolic blood pressure | 3 and 6 months
  Comparison of the diastolic blood pressure between enrolment, and 3 months and 6 months after enrolment
Evolution of the general clinical criteria : heart rate | 3 and 6 months
  Comparison of the heart rate between enrolment, and 3 months and 6 months after enrolment
Evaluation of the Rutherford score at enrolment and at 3 months and at 6 months after enrolment to estimate the clinical severity of venous insufficiency | 3 and 6 months
  Comparison of mean scores between enrolment and 3 months and 6 months after enrolment.
  The Rutherford questionnaire is the Venous Clinical Severity Score (VCSS) questionnaire without the compression part.
  The Rutherford questionnaire includes 9 hallmarks of venous disease, each scored on a severity scale from 0 to 3. In order to generate a dynamic score, the categories are scored individually, which adds emphasis to the most severe sequelae of venous disease that are likely to show the greatest response to therapy. These include skin changes and pigmentation, inflammation and induration, and ulcers (including number, size, and duration).
  Score from 0 to 27. A higher score means a worse outcome.
Evaluation of the use of care related or not to venous insufficiency 6 months post enrolment | 6 months
  Collection of medical events related or not to venous insufficiency (number of SAE, number of hospitalizations, number of medical and paramedical procedures)
Evaluation of compliance with the spa therapy | 3 weeks
  Comparison of the thermal treatments received by the patient during the spa therapy with the thermal treatments prescribed by the thermal doctor at the start of the spa therapy, collected in the spa treatment booklet
Evaluation of the specific quality of life by the WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) questionnaire | 3 and 6 months
  Quantitative improvement of the health status of all patients by comparison of the mean of Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) at baseline, 3 months and 6 months for all patients, and then only for patients with osteoarthritis
  The WOMAC is the validated index for the assessment of lower limb osteoarthritis according to a Likert scale with 5 possible answers (none = 0; minimal = 1; moderate = 2; severe = 3; extreme = 4) Scores from 0 to 100. A higher score means a worse outcome.
Comparison of the effictiveness of the treatment according to the limitation of the patient's walking (subgroup analysis according to patient mobility) | 6 months
  Comparison of the primary endpoint Chronic Venous Insufficiency specific Quality of life questionnaire (CIVIQ20) according to the limitation of the patient's walking (limitation of the walking is self reported by the patient)
  The 20-item questionnaire, which provides a global index and an outline of 4 quality-of-life dimensions-"pain" (4 items), "physical" (4 items), "psychological" (9 items), and "social" (3 items).
  Items on the CIVIQ-20 scale were scored from 1 to 5 which means a total score from 20 to 100.
  A higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Grenoble Alpes, Grenoble
  - Laboratoire TIMC, Grenoble

REFERENCES:
- [Background] Kim Y, Png CYM, Sumpio BJ, DeCarlo CS, Dua A. Defining the human and health care costs of chronic venous insufficiency. Semin Vasc Surg. 2021 Mar;34(1):59-64. doi: 10.1053/j.semvascsurg.2021.02.007. Epub 2021 Feb 3. PMID 33757637
- [Background] Carpentier PH, Blaise S, Satger B, Genty C, Rolland C, Roques C, Bosson JL. A multicenter randomized controlled trial evaluating balneotherapy in patients with advanced chronic venous insufficiency. J Vasc Surg. 2014 Feb;59(2):447-454.e1. doi: 10.1016/j.jvs.2013.08.002. Epub 2013 Oct 15. PMID 24135621
- [Background] Launois R. Health-related quality-of-life scales specific for chronic venous disorders of the lower limbs. J Vasc Surg Venous Lymphat Disord. 2015 Apr;3(2):219-27.e1-3. doi: 10.1016/j.jvsv.2014.08.005. Epub 2014 Oct 29. PMID 26993844
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- See also: [Anaes 1999] Evaluation et suivi de la douleur chronique chez l'adulte en médecine ambulatoire. Agence nationale d'accréditation et d'évaluation en santé. Recommandations et références professionnelles. Février 1999 — https://www.has-sante.fr/upload/docs/application/pdf/douleur1.pdf
- See also: [Queneau 2016] Press Therm Climat 2016;153:9-24 — https://www.academie-medecine.fr/wp-content/uploads/2016/10/Article-de-la-Presse-thermale.pdf